CLINICAL TRIAL: NCT06110130
Title: Effect of Empagliflozin on Podocyte Specific Proteins (Injury Markers) in African American Veterans With Non-Diabetic Chronic Kidney Disease
Brief Title: Effect of Empagliflozin on Podocyte Specific Proteins in African American Veterans With NDKD
Acronym: EMPA CKD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Sabyasachi Sen, MD, PhD, Chief of Endocrinology, Washington D.C. Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1770617
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Diseases
Keywords: Non-diabetic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Active Comparator): Placebo 10 mg orally daily
  Interventions: Drug: Placebo
- Empagliflozin (Active Comparator): Empagliflozin 10 mg orally daily
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Take Empagliflozin 10 mg orally daily for 4 months
  Arms: Empagliflozin
Drug: Placebo — Take Placebo 10 mg orally daily for 4 months
  Arms: Placebo

SUMMARY:
Primary Objective:To study podocyte specific injury markers in African American Veterans with non-diabetic kidney disease(NDKD), on empagliflozin therapy.

Primary Endpoint: Assess the effect of Empagliflozin on podocyte-specific proteins in exosomes isolated from subjects' urine, such as nephrin, podocalyxin and Wilms'Tumor (WT-1) protein.

Secondary Objective:

1. Correlate changes in exosome-based podocyte specific proteins with standardized biomarkers of kidney injury including urine albumin/creatinine ratio (ACR) and estimated GFR.
2. Correlate systemic inflammatory markers (focusing on vascular and endothelial function) that are already established such as interleukins (IL1, IL6, IL-12) , hs-CRP and arterial stiffness measures with urine exosome-based podocyte protein estimation.
3. Correlate urine podocyte-specific protein markers with APOL1 mRNA expression levels in blood mononuclear cells (MNC)

DETAILED DESCRIPTION:
Nephropathy is a progressive complication of DKD and NDKD and substantially increases morbidity and mortality. Clinicians frequently measure proteinuria using urine protein /creatinine and urine albumin/creatinine ratios, which in several instances do not manifest substantial improvement, even after an intervention such as SGLT2i, particularly if the intervention period is is less than 6 months. There is therefore a clear need for other markers of podocyte injury in early phases of chronic kidney disease.

Based on published studies, podocyte-specific injury proteins such as podocalyxin, Nephrin and Wilms tumor 1 (WT1) can be candidate marker proteins of injury. Urinary exosome analysis is a non-invasive and potentially more sensitive assay. These sensitive markers would reduce the need for biopsies to detect podocytopathy.

The Veterans Health Administration has been a prominent caregiver to the African American community across the United States. Over the past decade, investigators have established the basic population genetics and epidemiology of APOL1-associated kidney disease and are making progress in understanding disease mechanisms at the cellular and molecular levels. With therapeutic approaches for APOL1 kidney disease now being explored by many groups in pharma and academia, studies to assess the relationship of APOL1 gene expression levels with podocyte injury in CKD are of paramount importance and will better inform treatment in the near future. These studies may address one important cause of the significant racial disparity in CKD rates among African-Americans. This study aim to explore mechanistic insights gained from the effect of SGLT2i on podocyte injury markers further in the backdrop of APOL1 expression, to understand the potential therapeutic impact SGLT2i may have in this clinical context.

As APOL-1 gene mutation is much more common in African Americans and approximately 80% of VA population is African Americans, this study has been decided to enroll only from African American race in order to keep the population homogenous and achieve statistically significant results. Though the study will only include African Americans the study will be quite relevant in USA as worsening CKD is a major health problem in this country and the African American patient population is at particularly at a high risk for progressive CKD. A largely under-recognized public health issue, CKD is the ninth leading cause of death in the U.S. today. Although African Americans constitute 13% of the population, they suffer more than triple the rate of kidney failure of Caucasians.

ELIGIBILITY:
Inclusion Criteria:

1. African American veterans
2. Age > 18 years
3. eGFR ≥20-59 mL/min/1.73 m2 by the CKD-EPI equation, with or without any degree of albuminuria OR
4. eGFR 60-89, with UACR of ≥30mg/g
5. BMI = 18-39.9
6. Blood pressure controlled to ≤140/90
7. Subjects without diabetes: will be screened using routine glucose level test: of less than 126 fasting glucose or less than 200mg/dl of random or post glucose blood glucose level in standard of care laboratory workup.
8. Ability to provide informed consent before any trial related activities are conducted.

Exclusion Criteria:

1. Diagnosed with Type 1 or Type 2 Diabetes Mellitus
2. Any prescribed diabetes medication for patients, such as GLP1RA, SGLT2is, and sulphonylureas
3. If a patient is on statin, need to be on a stable dose for a month.
4. Biopsy proven diagnosis of glomerular disease/glomerulonephritis
5. Active smokers,
6. Active skin wounds undergoing treatment or recent surgery within 1 month (due to possible aberrations in glycemic control)
7. Women who are pregnant, planning to become pregnant, nursing mothers, women of childbearing potential not using birth control measure
8. Hypersensitivity to empagliflozin or any of the excipients in Jardiance, reactions such as angioedema
9. Patients on dialysis
10. eGFR less than 20 mL/min/1.73 m2 by the CKD-EPI equation
11. Planned surgery or planned hospital admission within 5 months of participation in the study
12. At the discretion of PI to ensure health, safety, and well-being of the veteran, participation in this study may be stopped (please see withdrawal criteria)
13. Patients with prior history of diagnosis of heart failure with documented EF of less than 50.
14. Proven diagnosis of Polycystic Kidney Disease.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To study kidney dysfunction and podocyte specific injury | 3 years
  To study kidney dysfunction and podocyte specific injury in African American Veterans with Non-diabetic kidney disease, following low dose of Empagliflozin therapy. Empagliflozin may be referred to as "Empa" hereafter. Correlate changes in exosome-based podocyte specific proteins with standardized biomarkers of kidney injury including urine albumin/creatinine ratio (ACR) and estimated GFR.

SECONDARY OUTCOMES:
Systemic inflammatory markers | 3 years
  Correlate systemic inflammatory markers (focusing on vascular function and endothelium) that are already established such as interleukins and hs-CRP and arterial stiffness with urine exosome-based podocyte protein estimation To correlate urine podocyte-specific protein markers and serum inflammatory markers with APOL1 mRNA expression levels in blood mononuclear cells (MNC) (c-kit positive cells)

CONTACTS AND LOCATIONS:
Overall Officials: Sabyasachi Sen, MD, Principal Investigator — Washington VA Medical Center
Locations (1):
- Washington DC Veterans Affairs Medical Center (688), Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No